CLINICAL TRIAL: NCT04476862
Title: Cerliponase Alfa Observational Study
Brief Title: Cerliponase Alfa Observational Study in the US
Status: Active, not recruiting | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 190-501
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Late-Infantile Neuronal Ceroid Lipofuscinosis Type 2
Keywords: Batten's Disease; CLN2; TPP1 enzyme
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses | interventions — cerliponase alfa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Cerliponase alfa patients: Patients who are currently on or plan to start taking cerliponase alfa within 60 days of signing the study informed consent form.
  Interventions: Drug: Cerliponase Alfa; Device: Administration Kit

INTERVENTIONS:
Drug: Cerliponase Alfa — Commercially available product provided to patient by participating clinic site.
  Other Names: Brineura
Device: Administration Kit — Commercially available administration kit provided to the patient by participating clinic site.

SUMMARY:
This is a multicenter, observational study for patients with a confirmed diagnosis of neuronal ceroid lipofuscinosis type 2 (CLN2 disease), also known as TPP1 deficiency, who intend to be or are currently being treated with cerliponase alfa. Patients receiving or expected to receive cerliponase alfa within 60 days of signing the informed consent form (ICF) may be eligible to enroll in the study, assuming all regulatory requirements for sites that have agreed to participate and protocol inclusion criteria are met. Data may be collected for all or some of the assessments as outlined in the protocol, dependent upon the clinic's and/or individual patient's standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with CLN2 disease.
2. Currently receiving or plan to begin treatment with cerliponase alfa.
3. Written informed consent/assent obtained.

Exclusion Criteria:

1. Currently receiving treatment in another investigational device or drug study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CLN2 patients who are currently taking or intend to take cerliponase alfa within 60 days of signing the informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2020-08-19 (Actual); Primary Completion 2030-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety surveillance of cerliponase alfa | 10 years
  To evaluate the long-term safety of cerliponase alfa in patients with neuronal ceroid lipofuscinosis Type 2 (CLN2 disease).

SECONDARY OUTCOMES:
Hypersensitivity | 10 years
  To further assess the occurrence of serious hypersensitivity reactions (including anaphylaxis), serious cardiovascular adverse events, and serious device-related complications.
Severe SAE impact on patient's motor and language functions | 10 years
  To evaluate the effects of Grade III or higher serious adverse events (SAEs) on patient performance on the CLN2 clinical rating scale (motor and language domains).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (16):
- United States (16):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Hospital, Washington D.C., District of Columbia
  - Advent Health, Orlando, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Boston Children's Hospital,, Boston, Massachusetts
  - Children's Hospital Minnesota, Minneapolis, Minnesota
  - NYU Langone Medical Center, New York, New York
  - Mt. Sinai School of Medicine, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No